CLINICAL TRIAL: NCT00005902
Title: A Prospective Natural History Study of VHL Patients With CNS Hemangioblastomas
Brief Title: Study of Brain and Spinal Cord Tumor Growth and Cyst Development in Patients With Von Hippel Lindau Disease
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000140; 00-N-0140
Record Dates: First submitted 2000-06-06; First posted 2000-06-07 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-05-08

CONDITIONS: Hemangioblastoma; Hippel Lindau Disease
Keywords: Brain; Brainstem; Cysts; Spinal Cord; MRI (Magnetic Resonance Imaging); Natural History
MeSH Terms: conditions — Hemangioblastoma; von Hippel-Lindau Disease; Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: 250 subjects with von Hippel-Lindau (VHL) disease.

SUMMARY:
The purpose of this study is to learn more about the growth of brain and spinal cord tumors and cysts that develop in association with them in patients with von Hippel-Lindau disease. It will examine how fast the tumors grow and try to determine what factors (for example, puberty , pregnancy, menopause, blood proteins, etc.) affect their growth.

Patients between the ages of 8 and 75 years who are enrolled in NIH s study of von Hippel-Lindau disease may be eligible for this 5-year study. Participants will have magnetic resonance imaging (MRI) of the brain and spinal cord and a thorough neurological history and examination at the start of the study. A blood sample will be taken for analysis of factors (hormones or other proteins) that may predict tumor growth. Follow-up clinic visits every 6 months will include a physical and neurological examination, blood tests, and MRI scans of the brain and spine. If symptoms or tumor growth requires more frequent follow-up, scans will be done at 3-month intervals.

Surgical removal of brain and spinal cord tumors is currently the treatment of choice when these lesions cause neurological problems. A better understanding of which tumors are likely to grow and which will remain stable may help guide physicians in treatment decisions and avoid unnecessary procedures.

DETAILED DESCRIPTION:
Hemangioblastomas of the cerebellum, brainstem, and spinal cord are frequent tumors in patients with von Hippel-Lindau (VHL) disease. Rarely, these lesions also affect the cerebrum. Patients often have multiple lesions, many of which are associated with cysts or syrinx. The current treatment for symptomatic lesions is surgical resection. Focused radiation is also being used in selected cases in an attempt to provide tumor control. The natural history of central nervous system (CNS) lesions in patients with VHL has not been addressed in a prospective study. It is not clear at which point these lesions will begin to grow, or develop cysts in the cerebellum or syrinx in the spinal cord, and systemic factors that influence tumor growth have not been identified. By identifying factors that predict or influence tumor progression or cyst development, we can more accurately recommend surgical or medical intervention at appropriate times and avoid unnecessary treatment for stable lesions. This natural experiment trial collected prospective radiological and clinical data on the growth of the central nervous system (CNS) hemangioblastomas and associated cysts. We prospectively collected information on systemic processes that may influence tumor progression, such as puberty, menopause, pregnancy, effects of hormone therapy, tumor load, serum erythropoietin level and hemoglobin/hematocrit levels.

This natural experiment trial has resulted in significant improvement in our understanding of the pathophysiology of VHL disease. Data from this trial have resulted in a better understanding of the origin and growth patterns of hemangioblastomas and endolymphatic sac tumors in patients with VHL disease. New therapies targeting hemangioblastomas in VHL disease are being devised based on information gathered from this study. We expect this natural experiment trial to continue to inspire new hypothesis-driven studies while improving the understanding and management of hemangioblastomas in VHL disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Ages 8-75.
  2. Confirmed diagnosis of von Hippel-Lindau disease.
  3. Presence of one or more cerebral, cerebellar or spinal cord hemangioblastomas on screening MRI.
  4. Able to give informed consent (or assent), or have a parent able to provide informed consent if a child.
  5. Karnofsky Performance Scale Score greater than or equal to 60.
  6. Have the capacity to undergo serial MRI scanning of the CNS without IV sedation.

EXCLUSION CRITERIA:

1. Clinically unstable condition.
2. Contraindication to MRI scanning such as surgery that involves metal clips or wires which might be expected to cause tissue damage or produce image artifacts.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll 250 subjects with von Hippel-Lindau (VHL) disease. Withdrawal/dropouts will not be replaced.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2001-02-15 (Actual)

PRIMARY OUTCOMES:
Determine the course of clinical and radiographic progression of VHL | Baseline, 12-24 month intervals
  The questions to be answered fall in the following general categories: 1. Course of Clinical Progression 2. Radiographic Progression 3. Post-treatment outcome (surgery and radiation) 4. Contributing factors 5. Genetic variability and effects on disease progression

SECONDARY OUTCOMES:
Determine the course of tumor and cyst growth after surgical and/or radiation intervention. | 12 24 months after surgery until withdrawal or death

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Chittiboina, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do plan to share IPD. we will share all IPD that results in a publication on a public repository, as required by most journals. the data will be de-identified and anonymized.

REFERENCES:
- [Derived] Lonser RR, Butman JA, Huntoon K, Asthagiri AR, Wu T, Bakhtian KD, Chew EY, Zhuang Z, Linehan WM, Oldfield EH. Prospective natural history study of central nervous system hemangioblastomas in von Hippel-Lindau disease. J Neurosurg. 2014 May;120(5):1055-62. doi: 10.3171/2014.1.JNS131431. Epub 2014 Feb 28. PMID 24579662
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-N-0140.html